CLINICAL TRIAL: NCT06388369
Title: A Randomized Phase I/II Study of Neoadjuvant Treatment With 177-Lutetium- PSMA-617 With or Without Ipilimumab in Subjects With Very High-risk Prostate Cancer Who Are Candidates for Radical Prostatectomy (NEPI Trial)
Brief Title: Neoadjuvant Lu-PSMA Radioligand Therapy and Ipilimumab in Men With Very High-risk Prostate Cancer
Acronym: NEPI
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Advanced Accelerator Applications (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-608
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Very High Risk Prostate Carcinoma
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Intervention Model Description: The first patients are enrolled - without randomization - into the Safety Cohort to assess whether the treatment regime under investigation, i.e. Ipilimumab (3mg/kg) + [177Lu]Lu-PSMA-617 RLT (7,4 GBq), is appropriately tolerated as per dose escalation algorithm.
  If it is established that Ipilimumab (3mg/kg) + [177Lu]Lu-PSMA-617 RLT (7,4 GBq) is appropriately tolerated, patients will be randomized into the two arms of the Analysis Cohort:
  * Arm A: Ipilimumab + [177Lu]Lu-PSMA-617 RLT
  * Arm B: [177Lu]Lu-PSMA-617 RLT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant Combination Therapy (Experimental): 4 cycles of Ipilimumab 3mg/kg + 2 cycles of 7,4 GBq [177Lu]Lu-PSMA-617
  Interventions: Radiation: [177Lu]Lu-PSMA-617; Drug: Ipilimumab
- Neoadjuvant Mono Therapy (Active Comparator): 2 cycles of 7,4 GBq [177Lu]Lu-PSMA-617
  Interventions: Radiation: [177Lu]Lu-PSMA-617

INTERVENTIONS:
Radiation: [177Lu]Lu-PSMA-617 — 2 cycles of 7,4 GBq [177Lu]Lu-PSMA-617 at 6 weeks intervals
Drug: Ipilimumab — 4 cycles of Ipilimumab 3mg/kg at 3 weeks intervals
  Arms: Neoadjuvant Combination Therapy

SUMMARY:
A randomized, open-label Phase I/II study of neoadjuvant treatment with [177Lu]Lu-PSMA-617 radioligandtherapy (LuPSMA) with or without Ipilimumab in participants with very high-risk prostate cancer who are candidates for Radical Prostatectomy.

DETAILED DESCRIPTION:
A randomized, open-label Phase I/II study of neoadjuvant treatment with [177Lu]Lu-PSMA-617 radioligandtherapy (LuPSMA) with or without Ipilimumab in participants with very high-risk prostate cancer who are candidates for Radical Prostatectomy.

The study will be initiated by a safety cohort regarding the [177Lu]Lu- PSMA-617 dose including 6 to 12 patients, who will receive combination therapy with [177Lu]Lu-PSMA-617 and Ipilimumab. The Safety-Run-In-Phase follows a "none of three or one of six patients experienced intolerable events" approach per dose level. That is: The first 3 patients will receive 4 courses of ipilimumab (3 mg/kg) and 2 courses of 3.7 GBq [177Lu]Lu-PSMA-617. If no more than one of these patients develop grade 4 adverse reactions (ARs) without recovery within 3 weeks, another 3 patients will receive the same dosage. If no grade 4 AEs are observed in this second set of patients, we will enroll an additional 3 patients to increase the [177Lu]LuPSMA 617 dose to 7.4 GBq. If no more than one of those patients develop grade 4 ARs without recovery within 3 weeks back to grade ≤1 or to baseline values, another 3 patients will receive the same increased dosage. Provided that these patients do not develop grade 4 ARs, randomization of patients will be started. If the "none of three or one of six patients experienced intolerable events" approach per dose level is not passed the study will be terminated at this point.

46 patients with newly diagnosed very high-risk prostate cancer will be randomly assigned in a 1:1 ratio (Ipilimumab + [177Lu]Lu-PSMA- 617 vs. [177Lu]Lu-PSMA-617 alone) to receive 2 cycles of 7,4 GBq [177Lu]Lu-PSMA-617 with or without 4 cycles of concomitant Ipilimumab 3mg/kg prior to prostatectomy. Radioligandtherapy will be given at 6 weeks intervals while ipilimumab will be given every 3 weeks. For application of ipilimumab and [177Lu]Lu-PSMA-617 within one cycle (week 1 and 7), [177Lu]Lu-PSMA-617 is administered on day 1 and ipilimumab on day 3. ADT will be applied to all patients during the neoadjuvant treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age
2. Signed an informed consent form (ICF) indicating that the participant understands the purpose of and procedures required for the study and is willing to participate in the study; participants must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
3. Histologically confirmed adenocarcinoma of the prostate including following criteria: Very High-risk defined by a total Gleason-Score ≥4+4 (ISUP-GG 4+5) and clinical stage cT3 (digital rectal examination or imaging based) plus clinical nodal status cN+ or Serum-PSA level >20ng/ml
4. Exclusion of metastases (M0) on conventional imaging and maximum oligometastatic status on PSMA PET imaging
5. Treatment naïve patients
6. Eastern Cooperative Oncology Group ECOG 0-1
7. Candidate for radical prostatectomy with pelvic lymph node dissection as per the investigator
8. Patients must be PSMA Positron Emission Tomography (PET) scan positive with a prostatic SUVmax > 12 (PRIMARY Score: 5) .
9. Following laboratory criteria must be obtained within 14 days prior to randomization:

   * Bone marrow reserve

     * White blood cells, WBC ≥ 2000/μL
     * Neutrophils ≥ 1500/μL
     * Platelets ≥ 100 x103/μL
     * Hemoglobin ≥ 9.0 g/dL
   * Hepatic:

     * AST/ALT ≤ 3 x ULN
     * Total Bilirubin ≤ 1.5 x ULN (except participants with Gilbert Syndrome, who may have total bilirubin < 3.0 mg/dL)
   * Renal:

     * Serum creatinine ≤ 1.5xULN
   * Endocrine:

     * TSH 0,4 - 4,0 mU/l = 0,4 - 4,0 μU/ml
     * If TSH is not in normal range, fT3 and fT4must be determined fT3 2,3 - 4,5 pg/ml = 3,5 -7,0 pmol/l fT4 0,8 - 1,8 ng/dl = 8 - 18 ng/l = 10 - 23 pmol/l
   * Albumin >3.0 g/dL (3.0 g/dL is equivalent to 30 g/L)
   * Electrolytes:

     * Potassium: 3.5-5 mmol/L
     * Sodium: 135-145 mmol/L
   * Pancreatic:

     * amylase, lipase ≤ 3 x ULN
   * alkaline phosphatase (range to be assessed in context of oligometastatic disease)
   * blood sugar < 200 mg/dL (11.1 mmol/L)
10. Sexually active patients must use a condom to prevent them from fathering a child and to prevent delivery of study treatment via seminal fluid to their partner for at least 14 weeks after the last dose of [177Lu]Lu-PSMA-617.
11. Tumor tissue of both prostate biopsy and radical prostatectomy specimen available for local histology review and reference pathology by Professor Henning Reis (Department of Pathology, University Hospital Frankfurt).

Exclusion Criteria:

1. Distant metastasis (clinical stage M1) on conventional imaging. Oligometastatic patients on exclusively PSMA PET imaging will not be excluded. Patients with PSA values below 20ng/ml and no evidence of nodal disease are excluded.
2. Prior treatment with androgen receptor antagonists. Treatment with GnRH analogs prior to ICF signature
3. Bilateral orchiectomy
4. History of prior systemic or local therapy for prostate cancer, including pelvic radiation for prostate cancer
5. Use of any investigational agent ≤4 weeks prior to randomization or any therapeutic procedure for prostate cancer at any time
6. Major surgery ≤4 weeks prior to randomization
7. Prior therapy with CTLA4 antibodies
8. Previous treatment with any of the following within 6 months of randomization:

   * Strontium-89, Samarium-153, Rhenium-186, Rhenium- 188, Radium-223,
   * Previous PSMA-targeted radioligand therapy
9. Any immunosuppressive therapy given within the past 30 days prior to study drug administration (excluding physiologic steroid hormone replacement and / or steroid therapy up to a maximum dose of 10 mg prednisone or equivalent per day)
10. Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy
11. Lack of availability for clinical follow-up assessments.
12. Other potential life-threatening malignancies within the past five years requiring treatment
13. Serious cardiac, gastrointestinal, hepatic or pulmonary disease reducing life expectancy to less than five years
14. Patients with serious intercurrent illness, requiring hospitalization.
15. Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders.
16. Patients carrying organ transplants and/or receiving continuous immunosuppressive medication (other than steroid therapy of up to 10 mg prednisone per day)
17. The patient is known to be positive for Human Immunodeficiency Virus (HIV) or other chronic infections (HBV, HCV) or has another confirmed or suspected immunosuppressive or immunodeficient condition.
18. Known hypersensitivity reaction to any of the components of study treatment
19. Known alcohol or drug abuse
20. Participation in another clinical study and use of any investigational or non-registered product (drug or vaccine) other than the study treatment within the 30 days before registration
21. Significant disease or condition which, in the investigator's opinion, would exclude the patient from the study
22. Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility to perform prostatectomy on time | During the intervention/procedure
  Feasibility will be defined as the ability to perform prostatectomy in at least 75% of the Analysis population 85 days after start of neoadjuvant treatment with a maximum delay by 3 weeks. A treatment arm will be deemed not feasible in the actual study if >25% of patients of that arm required a delay of surgery >3 weeks.
Clinical activity: Proportion of participants in the full analysis set who achieve a pCR | After surgery
  The proportion of participants in the full analysis set who achieve a pathological complete response (pCR). The assessment of pCR will be reviewed by the central pathologist for all randomized patients with Radical Prostatectomy with pelvic lymphadenectomy conducted. The proportion of participants in the full analysis set who achieve a MRD. The assessment of MRD will be reviewed by the central pathologist for all randomized patients with Radical Prostatectomy with pelvic lymphadenectomy conducted.

SECONDARY OUTCOMES:
Safety Profile of neoadjuvant treatment before radical prostatectomy | Start of neoadjuvant treatment up to 1 year after surgery
  Characterizing the safety profile of neoadjuvant treatment with Ipilimumab and [177Lu]Lu-PSMA-617 RLT before radical prostatectomy according to AEs and SAEs measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Safety Profile of neoadjuvant treatment before radical prostatectomy | Start of neoadjuvant treatment up to 1 year after surgery
  Measures of PSA progression-free survival for up to 1 year after prostatectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Clinic of Urology, Essen, Germany